CLINICAL TRIAL: NCT01991301
Title: The Safety and Efficacy of Carfilzomib -a Novel Proteasome Inhibitor- for the Prevention of Acute Graft Versus Host Disease
Brief Title: Carfilzomib for the Prevention of Graft Versus Host Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-12-9997-AN-CTIL
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Graft-versus-host Disease
Keywords: graft-versus-host disease; stem cell transplantation; matched unrelated donors; proteosmoe inhibitor; carfilzumib
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carfilzumib (Experimental): Carfilzomib at a dose of 20mg/m2 I.V. will be administrated at day 1, 2 post infusion of the stem cell (SC) graft to the first 10 patients. If no > grade II toxicity* the next 10 patients will receive Carfilzomib (27 mg/m2) at day 1,2 and 8, 9, 15 and 16. If no > grade II toxicity* the next 10 patients will receive 2-3 cycles of Carfilzomib (27 mg/m2) administered at day 1,2 8,9,15 and 16 post SC graft infusion.
  Interventions: Drug: carfilzumib

INTERVENTIONS:
Drug: carfilzumib — carfilzumib will be added to the standard regimen of drugs for prevention of graft-versus-host disease.

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of Carfilzumib, which is a novel biological agent used in the treatment of multiple myeloma in preventing graft-versus-host disease, after stem cells transplantation from unrelated donors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS/AML
2. 18 years or older and willing and able to comply with the protocol requirements.
3. LVEF ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
4. Patients undergoing 8-10/10 HLA matched unrelated and unmanipulated PBSC transplantation
5. Patients conditioned with reduced intensity or reduced toxicity conditioning i.e. Fludarabine combine with Treosulfan or 2-4 days of I.V Busulfan.
6. Patients must sign written informed consent.
7. Adequate birth control in fertile patients.

Exclusion Criteria:

1. Patients undergoing other type of transplantation or with other type of basic disease other than AML or MDS.
2. Patients with respiratory failure (DLCO < 30%).
3. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention.
4. Patients with > grade II liver renal toxicity.
5. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate
6. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
7. Creatinine > 2.0 mg/dl
8. ECOG-Performance status > 2
9. Uncontrolled infection
10. Pregnancy or lactation
11. CNS disease involvement
12. Pleural effusion or ascites > 1 liter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
incidence of acute graft-versus host disease | 3 months
  We will evaluate the incidence of acute GVHD, grading and organ involvementBY STANDARD INTERNATIONAL CRITERIA.

SECONDARY OUTCOMES:
incidence of chronic graft-versus-host disease | 1 year
  We will evaluate the progression of acute graft-versus-host disease to chronic graft-versus-host disease and the grading and organ involvement.
survival rate | 2 years
  We will evaluate overall and disease-free survival after stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Shimoni A, Shem-Tov N, Yerushalmi R, Danylesko I, Nagler A. Carfilzomib combined with cyclosporine and methotrexate for the prevention of graft-versus-host disease after allogeneic stem-cell transplantation from unrelated donors. Bone Marrow Transplant. 2021 Feb;56(2):451-456. doi: 10.1038/s41409-020-01044-5. Epub 2020 Sep 2. PMID 32873915